CLINICAL TRIAL: NCT06345144
Title: Learning Experience of Undergraduate Nursing Students in Pediatric Oncology Ward
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202307211RINC
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undergraduate nursing students

SUMMARY:
Clinical practices are crucial experiences for nursing students as they prepare themselves for future nursing work. Despite some research having been studied among Taiwanese nursing students in the past, there has been limited research into the experiences within pediatric oncology wards, where diseases are complex and frequently involve life-and-death issues. Therefore, the purpose of this study is to explore the experiences of undergraduate nursing students in pediatric oncology wards.

DETAILED DESCRIPTION:
Pediatric cancer is the leading cause of death in Taiwan for children aged 1-14. Despite advances in cancer diagnosis and treatment technology, pediatric cancer still requires highly professional and holistic health care. For healthcare professionals, it is a very challenging task. It can be assumed that for nursing students, the pressure of caring for children with cancer must be considerable. Additionally, pediatric care emphasizes family-centered care, meaning that during their clinical practices, nursing students not only need to learn skills related to caring for diseases but also understand the impact of cancer care on caregivers. This may lead to frustration or discouragement and potentially affecting their future careers in pediatric oncology wards Existing studies on nursing student clinical practice experiences in other wards have found that many nursing students have poor experiences due to insufficient technical skills, knowledge, and communication issues with both families and children. Therefore, utilizing qualitative research methods to understand nursing students' clinical practice experiences in pediatric oncology wards is crucial for identifying their learning needs and challenges. This study will involve in-depth interviews lasting for 30-60 minutes with nursing students who have completed their clinical practice in pediatric oncology wards, using semi-structured interview guides to elicit their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students in Taiwan
* Experienced clinical practice in pediatric oncology ward
* Who can describe their experiences in Chinese
* Understand and agree the purpose of this study

Exclusion Criteria:

* Not Undergraduate nursing students in Taiwan
* Haven't experienced clinical practice in pediatric oncology ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Undergraduate nursing students in Taiwan
  2. Experienced clinical practice in pediatric oncology ward
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Explore the experiences of undergraduate nursing students practicing in pediatric oncology wards. | up to 7 months
  With in-depth interviews lasting for 30-60 minutes with nursing students who have completed their clinical practice in pediatric oncology wards, using semi-structured interview guides to elicit their experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Wei-En Li, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No